CLINICAL TRIAL: NCT05110170
Title: A Multicenter, Randomized, Open-Label Phase Ⅲ Trial to Compare Efficacy and Safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01005) and ZOLADEX® in Patients With Breast Cancer
Brief Title: Efficacy and Safety of LY01005 in Patients With Breast Cancer Compared to ZOLADEX®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY01005/CT-CHN-303
Record Dates: First submitted 2021-11-03; First posted 2021-11-05 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; LY01005; Efficacy; Safety
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY01005 3.6 mg (Experimental): Intramuscular injections of LY01005 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: LY01005
- ZOLADEX® 3.6 mg (Active Comparator): Subcutaneous injections of ZOLADEX® 3.6 mg every 28 days for a maximum of 3 consecutive doses.
  Interventions: Drug: ZOLADEX® 3.6 mg

INTERVENTIONS:
Drug: LY01005 — LY01005 was administered as 3 intramuscular (IM) injections, 28 days apart. As concomitant medications, tamoxifen (10 mg/tablet, 1 tablet/time) was orally administered twice per day during the whole study period.
  Other Names: Goserelin Acetate Sustained-Release Microspheres for Injection
  Arms: LY01005 3.6 mg
Drug: ZOLADEX® 3.6 mg — ZOLADEX® was administered as 3 Subcutaneous (SC) injections, 28 days apart. As concomitant medications, tamoxifen (10 mg/tablet, 1 tablet/time) was orally administered twice per day during the whole study period.
  Other Names: Goserelin Acetate Implant 3.6 mg
  Arms: ZOLADEX® 3.6 mg

SUMMARY:
This is a multicenter, randomized, open-label, active comparator-controlled phase Ⅲ trial to compare efficacy and safety of Goserelin Acetate Sustained-Release Microspheres for Injection (LY01005) and ZOLADEX® in patients with breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active comparator-controlled phase Ⅲ trial using non-inferior design. A total of 188 patients with breast cancer who are suitable for endocrine therapy will be enrolled into the screening period from D-28 to D-1 before administration. Eligible subjects will be randomized in a 1:1 ratio to receive LY01005 3.6 mg intramuscularly or ZOLADEX ® 3.6 mg subcutaneously once every 28 days for three doses until intolerable toxicity, disease progression requiring other anti-tumor treatments, withdrawal of consent, loss to follow-up, death or the end of the whole study, and stratified according to history of chemotherapy (yes vs. no) and age (<45 vs. ≥45 years old). And all subjects will be also treated with tamoxifen orally twice per day (10 mg/tablet, 1 tablet/time). Blood samples will be collected at the specified time points of the study to detect serum E2, LH and FSH. Safety evaluation (including vital signs, physical examination, laboratory tests, 12 ECG, adverse events, etc.) will be conducted as required in the protocol. Additional blood samples will be collected from 12 subjects (PK subgroup) who are randomized to LY01005 group to assess the PK and PD characteristics of LY01005 in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 and <60 at screening, in pre-menopausal status defined as: (1) Menses within 1 year before enrolment; (2) Serum E2 >30 pg/mL and FSH ≤40 mIU/mL within 4 weeks before enrollment. (If patients received hysterectomy, they should only meet the second item.)
* Histologically confirmed ER+ primary breast cancer (ER+ defined as at least 10% of the cells examined by immunohistochemistry testing have estrogen receptors), TNM stage (according to the 8th edition of the AJCC Cancer Staging Manual): T1-T3, any N stage, M0 or Tis/T0, lymph node positive, M0.
* Patients who have previously received breast cancer-related surgery, have no known clinical residual local regional lesions after surgery (adjuvant radiotherapy was allowed after surgery), and are suitable for treatment with the combination of the study drug and tamoxifen as judged by the investigator (patients who have received neoadjuvant/adjuvant chemotherapy were allowed);
* Life expectancy of more than 9 months.
* ECOG score of ≤ 2.
* Female patients of child bearing potential who have a negative pregnancy test and their partners must agree to the use of non-hormonal contraception throughout the study period for at least 3 months after last dose.
* Patients who voluntarily sign an IRB-approved informed consent form before any trial-related activities, are willing to abide by the restrictions of the study, and complete the prescribed examinations.

Exclusion Criteria:

* Any evidence of distant metastatic lesions.
* Have received any neoadjuvant /adjuvant endocrine therapy for breast cancer previously.
* Have received a bilateral oophorectomy, ovarian radiotherapy, hypophysectomy or adrenalectomy, or who have pituitary lesions.
* Have received major surgery within 4 weeks prior to randomization.
* History or presence of another malignancy, other than surgically removed squamous/basal cell carcinoma of the skin or radically resected in situ cervical carcinoma, within the last 5 years.
* Presence of infectious diseases requiring intramuscular or intravenous drug therapy at the screening visit.
* Suffering from serious diseases within 6 months before the screening visit, including but not limited to: acute coronary syndrome, coronary revascularization, New York Heart Association (NYHA) class ≥ II cardiac insufficiency, severe unstable arrhythmia; Or the presence of fundus disease, severe osteoporosis, uncontrolled seizures, extensive bilateral lung disease diagnosed by high-resolution computed tomography, mental diseases that prevent the signing of informed consent at the screening visit.
* History of bleeding diathesis (i.e., disseminated intravascular coagulation [DIC] or clotting factor deficiency) or long-term anti-coagulant therapy (other than anti-platelet therapy).
* History of deep venous thrombosis, pulmonary embolism or stroke.
* Total bilirubin >1.5xULN, ALT or AST >2.5xULN, platelets <90 × 10^9/L, QTc interval >460ms, creatinine clearance < 30 mL/min (calculated according to Cockcroft-Gault formula) at the screening visit.
* Patients who are seropositive for hepatitis B surface antigen (HBsAg) must meet the following 2 conditions at the same time: 1. HBV DNA level: HBeAg-positive patients, HBV DNA ≥ 20,000 IU/ml [equivalent to 10^5 copies/mL]; HBeAg-negative patients, HBV DNA ≥ 2,000 IU/ml [equivalent to 10^4 copies/mL]; 2. ALT ≥ 2 x ULN).
* Patients who are seropositive for any one of hepatitis C virus antibody (HCV-Ab), human immunodeficiency virus antibody (HIV-Ab) or anti-treponema pallidum antibody (TP-Ab).
* Known to be allergic to the active ingredients or any excipients of GnRH analogues or tamoxifen.
* Unwilling to stop taking any drug that affects sex hormonal status.
* Have received any investigational drug, any investigational biological product or any investigational medical device, and discontinued within 1 month or 5 half-lives of the corresponding drug before the screening visit, whichever is longer.
* Female patients who are pregnant or breast-feeding.
* Other conditions considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 188 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of LY01005 compared with ZOLADEX®: the percentage of subjects with serum E2 maintaining at postmenopausal level (≤30 pg/mL) from Week 4 to Week 12 after the first dose. | from Week 4 to Week 12 after the first dose

SECONDARY OUTCOMES:
Incidence of adverse events (AE). | up to Week 12
Changes in serum E2 level after administration. | from baseline to Week 12
Changes in serum LH level after administration. | from baseline to Week 12
Changes in serum FSH level after administration. | from baseline to Week 12
PK subgroup: changes in serum E2 level after administration to assess PD characteristic of LY01005. | from baseline to Week 12
PK subgroup: changes in serum LH level after administration to assess PD characteristic of LY01005. | from baseline to Week 12
PK subgroup: changes in serum FSH level after administration to assess PD characteristic of LY01005. | from baseline to Week 12
PK subgroup: changes in serum goserelin level after administration to assess PK characteristic of LY01005. | from baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No